CLINICAL TRIAL: NCT06155370
Title: Construction of Gynecological Tumor Organoids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lei Li, professor, Peking Union Medical College Hospital
Other Study IDs: K4903 G&O organoids
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Gynecologic Cancer; Organoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biospecimen obtained from patients diagnosed with gynecological cancer from the cancer site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- cohort of cervical cancer organoids: organoids derived from cervical cancer
  Interventions: Other: construction of organoids from gynecological tumor
- cohort of endometrial cancer organoids: organoids derived from endometrial cancer
  Interventions: Other: construction of organoids from gynecological tumor
- cohort of ovarian cancer organoids: organoids derived from ovarian cancer
  Interventions: Other: construction of organoids from gynecological tumor
- cohort of vulva cancer organoids: organoids derived from vulva cancer
  Interventions: Other: construction of organoids from gynecological tumor
- cohort of vaginal cancer organoids: organoids derived from vaginal cancer
  Interventions: Other: construction of organoids from gynecological tumor
- cohort of gestational trophoblastic tumor organoids: organoids derived from gestational trophoblastic tumor
  Interventions: Other: construction of organoids from gynecological tumor

INTERVENTIONS:
Other: construction of organoids from gynecological tumor — organoids construction

SUMMARY:
This study focuses on the construction of a biological sample library for organoids and tumor tissues in gynecological tumors.

DETAILED DESCRIPTION:
Explore the construction and maintenance of a large-scale queue of gynecological tumor organoids. Beijing Daxiang Technology Co., Ltd. provides corresponding technical support and chip design. Gynecological oncology center provides tumor samples, clinical information, and pathological support, and biological sample library provides technical support, storage space, and quality management.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 or older, an informed consent form is provided;
2. The preoperative tumor burden assessment and intraoperative researcher team believe that sampling is feasible;
3. Having relevant requirements for sample library storage;
4. Surgical treatment at Peking Union Medical College Hospital.

Exclusion Criteria:

1. Unable to meet all inclusion criteria;
2. The research team considers any situations or considerations that may hinder normal pathological assessment.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Those diagnosed with gynecological oncology, including cervical cancer, endometrial cancer, ovarian cancer, vulva cancer, vaginal cancer, and gestational trophoblastic tumor.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Construction of BioBank | one year
  BioBank including organoids banks, tissue banks, PDX banks, immune cell banks, and primary banks from other tissue sources

SECONDARY OUTCOMES:
Drug sensitivity detection based on organoids banks | one year
  Exploring drug sensitivity detection in gynecological tumors based on organoid libraries
Exploring the molecular mechanism based on organoids banks | one year
  Exploring the molecular mechanism of gynecological tumor pathogenesis based on organoid banks